CLINICAL TRIAL: NCT02232477
Title: An Extension Study of Intrathecal Enzyme Replacement for Cognitive Decline in Mucopolysaccharidosis I
Brief Title: Extension Study of Intrathecal Enzyme Replacement for Cognitive Decline in MPS I
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Termination of study by investigator related to COVID pandemic.
Sponsor: agnes chen (Other)
Collaborators: University of Minnesota (Other); UCSF Benioff Children's Hospital Oakland (Other); University of California, Los Angeles (Other); The Ryan Foundation (Other); Rare Diseases Clinical Research Network (Network); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, agnes chen, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Organization: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRC-002 (100)
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Results first posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Mucopolysaccharidosis I; Cognitive Decline
MeSH Terms: conditions — Mucopolysaccharidosis I; Cognitive Dysfunction | interventions — Iduronidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open-label treatment (Experimental): laronidase 1.74 mg IT q 3 months for five years
  Interventions: Drug: Intrathecal recombinant human alpha iduronidase

INTERVENTIONS:
Drug: Intrathecal recombinant human alpha iduronidase — Intrathecal recombinant human alpha iduronidase every 3 months
  Other Names: Aldurazyme

SUMMARY:
This is a five-year extension study of the pilot study, "Intrathecal Enzyme Replacement for Cognitive Decline in MPS I". Participants must have completed the pilot study to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has completed the MIRC-002 study of intrathecal enzyme replacement therapy for cognitive decline in mucopolysaccharidosis I
2. Age six years or older.
3. Subject and/or guardian willing and able to provide written informed consent.
4. Negative urine pregnancy test at screening (non-sterile females of child-bearing potential only)
5. Currently using two acceptable methods of birth control as determined by the investigator and willing to continue to use acceptable birth control during their participation in the study (non-sterile females of child-bearing potential who are sexually active only)
6. Willing and able to comply with study procedures. For example, the subjects must be able to complete written and computer-based testing. The subjects must be able to lie still in the MRI scanner for at least 40 minutes without sedation.

Exclusion Criteria:

1. The subject has undergone hematopoietic stem cell transplantation
2. Recent initiation of intravenous Aldurazyme® therapy with less than 6 months of therapy. Subjects who have been receiving Aldurazyme® therapy for more than 6 months, and those who have never received Aldurazyme® therapy, will be allowed to enroll
3. Pregnant or lactating, or considering pregnancy
4. Receipt of an investigational drug or procedure other than intrathecal Aldurazyme® within 30 days of enrollment
5. A condition, medical or other, that prevents participation in the study, including severe auditory or visual impairment, significant lumbar pathology, lumbar catheter, or recent major surgery within 6 weeks that would preclude their ability to participate.
6. Infusion reactions to intravenous or intrathecal Aldurazyme® therapy that are life-threatening or require emergent intervention such as epinephrine, cardiopulmonary resuscitation, or hospitalization
7. The subject has severely impaired spinal CSF flow, demonstrated by failure of appearance of radionuclide in the basal cisterns by 4 hours after intra-lumbar administration.
8. The subject has a coagulopathy, as identified by a platelet count of less than 50,000, an INR of 1.5 or greater, or a PTT that is 1.5 times the upper limit of normal for the laboratory from which it was drawn.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-label Treatment
Started | 6
Completed | 4
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.33 (3.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: Hopkins Verbal Learning Test
Description: Mean intra-subject change in total recall score on the Hopkins Verbal Learning Test between baseline/screening for MIRC-002 and the subject's final visit.
  The Hopkins Verbal Learning Test measures verbal memory. The subject is read a list of words and asked to memorize as many words as possible. The scale ranges from 0 to 36, with higher scores indicating a better outcome.
  Two relevant time points: Baseline and the subject's final visit. Because this study ended prematurely for due to the pandemic, the subject's final visit was at the 12-month time point for one subject, 24-months for one subject, 36-months for two subjects, and 48-months for two subjects.
  Calculation: The total recall score at Baseline was subtracted from the total recall score at the subject's final visit and mean change and standard deviation were reported.
Time Frame: zero to 48 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open-label Treatment
Number analyzed (Participants) | 6
score on a scale | -1.67 (2.58)

ADVERSE EVENTS:
Time Frame: 5 years, 6 months
Arm/Group | Open-label Treatment
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Treatment (N=6)
headache (Nervous system disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (4)
corneal transplant (Eye disorders) | 1 (1)
spinal cord injury (Nervous system disorders) | 1 (1)
psychiatric symptoms (Psychiatric disorders) | 1 (1)
hydrocephalus (Nervous system disorders) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 1 (1)
VP shunt infection (Nervous system disorders) | 1 (1)
small bowel obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Treatment (N=6)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (3)
mitral valve disease (Cardiac disorders) | 1 (1)
anxiety (Psychiatric disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 4 (18)
stress fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
glaucoma (Eye disorders) | 1 (1)
corneal transplant (Eye disorders) | 1 (1)
blurred vision (Eye disorders) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
aphthous ulcer (General disorders) | 1 (1)
urinary incontinence (Renal and urinary disorders) | 1 (1)
sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
otitis media (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT02232477/Prot_SAP_000.pdf